CLINICAL TRIAL: NCT06632431
Title: Clinicopathological Analysis of Endometrial Carcinoma in the View of Old and New International Federation of Gynecology and Obestetrics (FIGO)
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, yousra hassanin abdelghafour, Demonstrator of Pathology, Faculty of Medicine , Assiut University, Assiut, Egypt, Assiut University
Other Study IDs: 04-2024-200910
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Clinicopathological; Endometrial Carcinoma; Federation of Gynecology and Obestetrics
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial cancer group: Patients diagnosed with endometrial cancer (EC) who underwent surgical staging (total hysterectomy and bilateral salpingo-oophorectomy)
  Interventions: Other: Endometrial cancer (EC)

INTERVENTIONS:
Other: Endometrial cancer (EC) — Endometrial cancer (EC) who underwent surgical staging (total hysterectomy and bilateral salpingo-oophorectomy) Histopathological slides for these cases will be reexamined and staged according to both the Federation of Gynecology and Obestetrics (FIGO) 2009 and updated Federation of Gynecology and Obestetrics (FIGO) 2023 endometrial staging systems. Upstaging refers to reclassification to a higher stage in the FIGO 2023 system compared to Federation of Gynecology and Obestetrics (FIGO)2009, while downstaging is the opposite.
  All patients underwent lymph node dissection except those with Stage IA-Grades I and II endometrioid endometrial cancer and tumor size <2 cm.

SUMMARY:
Assess the percentage change in stage and risk stratification for patients with endometrial cancer when transitioning from the FIGO 2009 endometrial staging system to the updated FIGO 2023 endometrial staging system.

Investigate the prognostic impact of the FIGO 2023 endometrial staging system on patient survival.

Evaluate how the shift in stage classification between the FIGO 2009 and FIGO 2023 systems influences adjuvant management decisions for endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer is the commonest gynecological cancer mostly affecting women in the post-menopausal age group . The average age of women diagnosed with endometrial cancer is 60. It's uncommon in women under the age of 45. The vast majority of endometrial cancers are carcinomas (usually adenocarcinomas). The five-year survival rate for endometrial adenocarcinoma following appropriate treatment is 80%. More than 70% of women diagnosed have Federation of Gynecology and Obestetrics (FIGO) stage I cancer, which has the best prognosis. Stage III and especially Stage IV cancers has a worse prognosis, but these are relatively rare, occurring in only 13% of cases. The median survival time for stage III-IV endometrial cancer is nine to ten months.

The FIGO 2023 staging system provides a refined framework for managing endometrial cancer, benefiting patient care and outcomes as the FIGO 2023 staging system for endometrial cancer offers several advantages over the previous FIGO 2009 system

1. Improved Prognostic Prediction: The 2023 system predicts survival more accurately, validated by five studies and It adds granularity to prognostic assessment, identifying treatment-relevant subgroups of patients.
2. Incorporation of Molecular Measures as The 2023 system integrates molecular parameters, reflecting their impact on prognosis (similar to breast cancer staging)
3. Risk Stratification: It incorporates risk stratification, aiding better prognosis definition and treatment decisions.
4. Enhanced Understanding of Endometrial Carcinomas: The 2023 system clarifies the diverse biological nature of endometrial cancers, allowing for better-adapted treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with endometrial cancer (EC) who underwent surgical staging (total hysterectomy and bilateral salpingo-oophorectomy) between January 1, 2018, and December 31, 2022 with available medical records since diagnosis and at least follow up 2 years and received adjuvant treatment and available histopathological slides and blocks.

Exclusion Criteria:

- Patients who received neoadjuvant chemotherapy, had recurrent endometrial cancer, had multiple cancers, lacked histopathological slides and formalin-fixed paraffin-embedded blocks or lacked medical records were excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women will be clinicopathological analysis of endometrial carcinoma
Study Population: Patients diagnosed with endometrial cancer (EC) who underwent surgical staging (total hysterectomy and bilateral salpingo-oophorectomy) between January 1, 2018, and December 31, 2022 with available medical records since diagnosis and at least follow up 2 years and received adjuvant treatment and available histopathological slides and blocks.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in stage | One years after the start of study
  Percentage change in stage will be recorded for patients with endometrial cancer when transitioning from the FIGO 2009 endometrial staging system to the updated FIGO 2023 endometrial staging system.

SECONDARY OUTCOMES:
Risk stratification | One years after the start of study
  Risk stratification will be recorded for patients with endometrial cancer when transitioning from the FIGO 2009 endometrial staging system to the updated FIGO 2023 endometrial staging system.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.